CLINICAL TRIAL: NCT00085800
Title: Dietary Fiber and Cardiovascular Inflammatory Markers
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1255; R01HL076271 (NIH); NCT00294138 (obsolete NCT alias)
Record Dates: First submitted 2004-06-14; First posted 2004-06-17 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2008-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Non-insulin Dependent; Hypertension; Obesity; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Type 2; Hypertension; Obesity; Inflammation

SUMMARY:
To investigate the relationship between dietary fiber and cardiovascular inflammatory markers.

DETAILED DESCRIPTION:
BACKGROUND:

Recent studies have found that diets with higher fiber intake are associated with a reduction in cardiovascular disease (CVD). However, the association does not prove that dietary fiber is actually responsible for lower CVD risk nor does it illuminate potential mechanisms of lower risk if present. Since the diet-CVD connection is strong, and given that CVD is a major contributor to morbidity and mortality, additional information would be valuable. Our preliminary studies and the work of others suggest that there is a significant association between C-reactive protein (CRP) and dietary fiber intake. These observations led us to the following unifying hypothesis: Diets high in fiber are associated with lower levels of inflammatory markers. Our long-term goal is to determine whether inflammation is a key mediator in the link between fiber intake and cardiovascular disease risk.

DESIGN NARRATIVE:

The three specific aims of the project are 1: To determine whether total dietary fiber and or fiber supplementation is associated with levels of inflammatory markers (CRP, fibrinogen, WBC) among adult participants with obesity, hypertension, or diabetes in the National Health and Nutrition Examination Survey 1999-2000; 2: To determine whether 3 weeks on a diet naturally high in fiber (30g/day), or on a diet high in fiber through supplementation, will significantly reduce inflammatory markers compared to a diet low in fiber, in a clinical trial among 30 lean and 30 obese adult hypertensive volunteers; and 3: To determine whether 3 months on a diet supplemented with moderate fiber (extra 7g/day), or high fiber (15g/day), will significantly reduce inflammatory markers compared to a usual diet low in fiber (average 10-15g/day) in a three-month long clinical trial among 180 obese adult volunteers.

To accomplish these aims, three related studies will be conducted. The first will utilize existing data contained in the National Health and Nutrition Examination Survey, a national database of 5773 non-institutionalized adults. The second study will be an additional procedure and laboratory examination to an existing R01 by one of the investigators, to examine the impact of a diet naturally high in fiber on CRP and other inflammatory markers. The third study will consist of new primary data collection in 180 volunteers to evaluate the effect of different levels of fiber supplementation on CRP, fibrinogen, WBC, and interleukin-6. By using existing data, taking advantage of an ongoing protocol, and adding new information through primary data collection, the investigators hope to dramatically increase their understanding of the association between dietary fiber and cardiovascular inflammatory markers. This information could serve to guide constructive changes in nutritional guidelines for reducing CVD risk for millions of at-risk individuals.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana King — Medical University of South Carolina